CLINICAL TRIAL: NCT02756520
Title: Characterisation of Patient Profile and Contemporary Treatment of Pre-dialytic Chronic Kidney Disease (CKD) in Patients Receiving a Restricted Protein Diet Supplemented With Ketosteril® - a Drug Utilisation Study (DUS)
Brief Title: Observational Study on CKD Treatment With a Ketosteril Supplemented Protein-restricted Diet (Keto-024-CNI)
Status: Completed | Type: Observational
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Other Study IDs: Keto-024-CNI
Record Dates: First submitted 2016-04-27; First posted 2016-04-29 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease, pre-dialytic; Ketosteril, keto-acids; diet, protein-restricted; renal function
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic kidney disease (pre-dialysis): Observational study: supplemented protein-restricted diet
  Interventions: Other: Observational study: Supplemented protein-restricted diet

INTERVENTIONS:
Other: Observational study: Supplemented protein-restricted diet — Observational study: Supplemented protein-restricted diet

SUMMARY:
The purpose of this study is to characterize the patient and disease profile under the influence of a protein-restricted diet supplemented with keto acids/amino acids (KA/AA), focusing on the progression of chronic renal insufficiency, calcium and phosphorus metabolism, nutritional status, patient compliance to diet and Ketosteril intake as well as the persistent dietary education to ensure compliance in a large group of pre-dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* non-dialyzed patients with CKD
* indication for Ketosteril according to package insert (PI), including a glomerular filtration rate (GFR) < 25 mL/min
* accepted supplemented protein-restricted diet and newly starting with Ketosteril (treatment naïve, i.e., never treated with Ketosteril before)
* adult patients ≥ 18 years

Exclusion Criteria:

* active cancer diseases
* pregnancy or breast feeding
* hypersensitivity to active substances or to any of the excipients in Ketosteril
* hypercalcaemia
* major disorder of amino acid metabolism, e.g., hereditary diseases
* participation in any clinical trial with an investigational drug within 30 days prior to start of study or during the study
* illiteracy or incapability to read or write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pre-dialytic chronic kidney disease patients treated at nephrology units of selected hospitals in China
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Patient compliance to Ketosteril (number of tablets taken; patient reported) | 12 months
  This is an observational study aiming to characterise the patient profile and contemporary treatment of pre-dialytic chronic kidney disease (CKD) in patients receiving a restricted protein diet supplemented with Ketosteril®. There is no distinction between primary and secondary outcome measures in the observational plan, and only Routine procedures are documented.
  Patient compliance to Ketosteril will be assessed daily, for a total of 12 months.

SECONDARY OUTCOMES:
Patient compliance to diet (protein and energy intake; investigator and patient-reported, based on patient diary and a routine 3-day food diary) | Monthly, starting 1 month after enrolment, for a total of 12 months
  This is an observational study aiming to characterise the patient profile and contemporary treatment of pre-dialytic chronic kidney disease (CKD) in patients receiving a restricted protein diet supplemented with Ketosteril®. There is no distinction between primary and secondary outcome measures in the observational plan, and only Routine procedures are documented.
CKD stage (according to Kidney Disease Improving Global Outcomes [KDIGO] guideline) | At baseline and 3, 6, 9 and 12 months after enrolment
Presence of comorbidities | At baseline
Serum creatinine | At baseline and 3, 6, 9 and 12 months after enrolment
24h urinary protein | At baseline and 3, 6, 9 and 12 months after enrolment
Urinary microalbumin | At baseline and 3, 6, 9 and 12 months after enrolment
Serum urea | At baseline and 3, 6, 9 and 12 months after enrolment
Creatinine clearance | At baseline and 3, 6, 9 and 12 months after enrolment
Glomerular Filtration Rate (GFR) | At baseline and 3, 6, 9 and 12 months after enrolment
Estimated GFR (eGFR) | At baseline and 3, 6, 9 and 12 months after enrolment
Fasting blood glucose | At baseline and 3, 6, 9 and 12 months after enrolment
Fasting plasma glucose | At baseline and 3, 6, 9 and 12 months after enrolment
Haemoglobin A1c (HbA1c) | At baseline and 3, 6, 9 and 12 months after enrolment
Serum triglyceride | At baseline and 3, 6, 9 and 12 months after enrolment
Serum cholesterol | At baseline and 3, 6, 9 and 12 months after enrolment
Serum high-density lipoprotein (HDL) | At baseline and 3, 6, 9 and 12 months after enrolment
Serum low-density lipoprotein (LDL) | At baseline and 3, 6, 9 and 12 months after enrolment
Serum calcium | At baseline and 3, 6, 9 and 12 months after enrolment
Serum phosphate | At baseline and 3, 6, 9 and 12 months after enrolment
Serum parathyroid hormone (PTH) | At baseline and 3, 6, 9 and 12 months after enrolment
Body weight | At baseline and 3, 6, 9 and 12 months after enrolment
Skinfold thickness | At baseline and 3, 6, 9 and 12 months after enrolment
Serum total protein | At baseline and 3, 6, 9 and 12 months after enrolment
Serum albumin | At baseline and 3, 6, 9 and 12 months after enrolment
Serum prealbumin | At baseline and 3, 6, 9 and 12 months after enrolment
Body mass index (BMI) | At baseline and 3, 6, 9 and 12 months after enrolment
Subjective global assessment (SGA) | At baseline and 3, 6, 9 and 12 months after enrolment
Decline in eGFR | At 3, 6, 9 and 12 months after enrolment
Worsening of CKD stage | At 3, 6, 9 and 12 months after enrolment
Start of dialysis | At 3, 6, 9 and 12 months after enrolment
Presence of a 50% reduction in eGFR | At 3, 6, 9 and 12 months after enrolment
Serum bicarbonate | At baseline and 3, 6 and 12 months after enrolment
Serum haemoglobin | At baseline and 3, 6 and 12 months after enrolment
Serum potassium | At baseline and 3, 6 and 12 months after enrolment
Reported nausea and vomiting | At baseline and 3, 6 and 12 months after enrolment
Presence of concomitant disease | At 3, 6, 9 and 12 months after enrolment
Administration of concomitant medication | At 3, 6, 9 and 12 months after enrolment
Discontinuation of diet and Ketosteril with the reasons for discontinuation as reported by the investigator | Monthly starting at 1 month after enrolment for up to 12 months
Acceptance of diet as documented in the patient diary | Daily for up to 12 months
Appetite change as documented in the patient diary | Daily for up to 12 months
Change of food intake as documented in the patient diary | Daily for up to 12 months
Adverse events including adverse drug reactions and serious adverse events | At 3, 6, 9 and 12 months after enrolment
Blood pressure | At baseline and 3, 6, 9 and at 12 months after enrolment
Heart rate | At baseline and 3, 6, 9 and at 12 months after enrolment
Body temperature | At baseline and 3, 6, 9 and at 12 months after enrolment

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Xiangmei, Beijing, Beijing Municipality, China